CLINICAL TRIAL: NCT07026149
Title: Perioperative Treatment of Combined Radiotherapy With SOX, Apatinib and Camrelizumab for Resectable Locally Advanced Gastric or Esophagogastric Junction Adenocarcinoma: A Phase II Trial
Brief Title: Perioperative Treatment of Combined Radiotherapy With SOX, Apatinib and Camrelizumab for Oesophagogastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024373
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Gastric and Gastroesophageal Junction (GEJ) Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Radiotherapy and Apatinib and Camrelizumab and S-1 and Oxaliplatin
  Interventions: Drug: Apatinib+Camrelizumab+SOX; Radiation: Preoperative Radiotherapy

INTERVENTIONS:
Drug: Apatinib+Camrelizumab+SOX — Apatinib 250mg+Camrelizumab 200mg +S-1, Oxaliplatin, q3w
Radiation: Preoperative Radiotherapy — Radiotherapy was administered using IMPT or IMRT. The target volume includes the gastric lesion, and regional lymph nodes. A regimen of 41.4 Gy in 23 fractions is preferred.

SUMMARY:
The study is being conducted to evaluate the efficacy, safety and tolerability of radiotherapy and chemotherapy, apatinib with camrelizumab in the neoadjuvant (prior to surgery) and adjuvant (after surgery) treatment of previously untreated adults with gastric and gastroesophageal junction (GEJ) adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Has previously untreated localized gastric or GEJ adenocarcinoma as defined by T3-4N+M0;
* Plans to proceed to surgery following pre-operative chemotherapy. Has an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1.
* Has adequate organ function.
* Male participants of childbearing potential must agree to use an adequate method of contraception for the course of the study through 120 days after the last dose of therapy.
* Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of therapy.
* Has life expectancy of greater than 12 months.

Exclusion Criteria:

* Uncontrolled hypertension ( systolic ≥140 mmHg or diastolic ≥90 mmHg despite antihypertensive therapy)
* Known hypersensitivity to any of the study drugs or excipients.
* Known hereditary or acquired bleeding and thrombotic tendencies (e.g. hemophiliacs, coagulation disorders, thrombocytopenia, etc.);
* Congenital or acquired immune deficiency (e.g. HIV infected)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-08 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response | Up to 6 weeks after completion of radiotherapy and 3 cycles (each cycle is 21 days) of neoadjuvant drug treatment

SECONDARY OUTCOMES:
Total Pathological Complete Response (tpCR) | Up to 6 weeks after completion of radiotherapy and 3 cycles (each cycle is 21 days) of neoadjuvant drug treatment
Major pathological response(MPR) | Up to 6 weeks after completion of radiotherapy and 3 cycles (each cycle is 21 days) of neoadjuvant drug treatment
Margin-free (R0) resection rate | Up to 6 weeks after completion of radiotherapy and 3 cycles (each cycle is 21 days) of neoadjuvant drug treatment
Lymph node status after neoadjuvant therapy (ypN staging) | Up to 6 weeks after completion of radiotherapy and 3 cycles (each cycle is 21 days) of neoadjuvant drug treatment
DFS | up to 2 years
OS | up to 2 years
Local control rate | up to 2 years
AEs | Up to approximately 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Li C, Tian Y, Zheng Y, Yuan F, Shi Z, Yang L, Chen H, Jiang L, Wang X, Zhao P, Zhang B, Wang Z, Zhao Q, Dong J, Lian C, Xu S, Zhang A, Zheng Z, Wang K, Dang C, Wu D, Chen J, Xue Y, Liang B, Cheng X, Wang Q, Chen L, Xia T, Liu H, Xu D, Zhuang J, Wu T, Zhao X, Wu W, Wang H, Peng J, Hou Z, Zheng R, Chen Y, Yin K, Zhu Z. Pathologic Response of Phase III Study: Perioperative Camrelizumab Plus Rivoceranib and Chemotherapy Versus Chemotherapy for Locally Advanced Gastric Cancer (DRAGON IV/CAP 05). J Clin Oncol. 2025 Feb;43(4):464-474. doi: 10.1200/JCO.24.00795. Epub 2024 Oct 9. PMID 39383487